CLINICAL TRIAL: NCT06000657
Title: Efficacy and Safety of Switching to Vemliver (Tenofovir Alafenamide) From Entecavir in Chronic Hepatitis B: A Multi-Center, Phase IV, Open-Label, Randomized, Active-Controlled, Non-Inferiority Trial.
Brief Title: Efficacy and Safety of Switching to Vemliver From Entecavir in Chronic Hepatitis B Patients Previously Treated With Entecavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DWVMLV_P401
Record Dates: First submitted 2023-07-16; First posted 2023-08-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Chronic Hepatitis B patients who pretreated with Entecavir
  Interventions: Drug: Vemliver tablet
- Comparator group (Active Comparator): Chronic Hepatitis B patients who pretreated with Entecavir
  Interventions: Drug: Baracross Tablet

INTERVENTIONS:
Drug: Vemliver tablet — Chronic Hepatitis B Patients Who Pretreated with Entecavir switching to Vemliver tab (Tenofovir Alafenamide Hemitartrate)
  Arms: Treatment group
Drug: Baracross Tablet — Chronic Hepatitis B Patients Who Pretreated with Entecavir continuting treatement with Baracross Tablet
  Arms: Comparator group

SUMMARY:
Enroll patients who are pre-treated with Entecavir at least 24 weeks and confirmed HBV antiviral (HBV DNA <69 IU/mL) effects.

Subjects are given one test drug or comparator once a day for 48 weeks according to the results of random assignments, and their HBV antiviral inhibitory effect and safety are evaluated at 24 and 48 weeks visits.

DETAILED DESCRIPTION:
Enroll patients who are pre-treated with Entecavir at least 24 weeks and confirmed HBV antiviral (HBV DNA <69 IU/mL) effects.

At the time of screening, potential test subjects of this test are selected by retrospectively collecting information on disease status and prognosis-related factors, including ETV administration information, among those who voluntarily agreed to participate in this clinical trial.

HBeAg status (positive vs. positive) through Visit 1's Heptatis B Serology test before administering clinical trial drugs to test subjects who finally qualify for selection/exclusion criteria at the baseline. Voice) is set as a stratification factor and is randomly assigned to each test institution.

Subjects are given one test drug or comparator once a day for 48 weeks according to the results of random assignments, and their HBV antiviral inhibitory effect and safety are evaluated at 24 and 48 weeks visits.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 19 years and older as of the date of written consent.
2. Individuals with a positive HBsAg for at least 24 weeks prior to screening or a history of chronic hepatitis B.
3. Individuals with chronic hepatitis B who have been receiving ETV 0.5 mg as monotherapy for at least 24 weeks and have expressed the intention to switch to Barakros tablets or Bemeliver tablets.
4. Participants with good adherence to ETV 0.5 mg monotherapy confirmed through questionnaire (≥80%).
5. Participants who have demonstrated viral suppression efficacy (HBV DNA <69 IU/mL) and are deemed to require monotherapy with Tenofovir alafenamide or ETV for at least 48 weeks.
6. Individuals who voluntarily agree to participate in the clinical trial and have signed the informed consent form.

   Exclusion Criteria:

   Medical history or surgical (treatment) history at the time of screening visit:

   ① Individuals diagnosed with substance abuse or alcohol addiction within the past year of screening.
   * Confirmed diagnosis of malignant tumors, including liver cancer, within the past 5 years.

     * Organ or bone marrow transplant recipients.

   Coexisting conditions at the time of screening visit:

   ① Non-selective clinical signs/symptoms in non-selective liver disease.
   * Galactose intolerance, lactase deficiency, or glucose-galactose malabsorption.

     * Kidney disease patients requiring hemodialysis or peritoneal dialysis. ④ Other clinically significant cardiovascular, respiratory, neurological, or psychiatric conditions considered inappropriate for participation in the clinical trial according to the participant's judgment.

   Laboratory test results at the time of screening visit:

   ① Co-infection with HCV and HIV.
   * Hemoglobin <8 g/dL.

     * Impaired renal function. ④ ALT >3 × ULN.

   Anticipated use of the following drugs during the specified period:

   During the clinical trial period:
   * Immunosuppressants.

     * Systemic corticosteroids administered at a dose equal to or greater than a restricted dose for more than 2 weeks.

       * Drugs affecting renal excretion, drugs with renal or hepatic toxicity. ④ Anti-HBV drugs other than investigational medicinal products. ⑤ Hepatotonics.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
HBV viral suppression rate | 48 weeks
  HBV viral suppression rate at 48 weeks post-baseline

SECONDARY OUTCOMES:
HBV viral suppression rate | 24 weeks
  HBV viral suppression rate at 24 weeks post-baseline
ALT normalization rate | 24 weeks
  ALT normalization rate at 24 weeks post-baseline
ALT normalization rate | 48 weeks
  ALT normalization rate at 48 weeks post-baseline
Change from baseline in ALT | 24 weeks
  Change from baseline in ALT at 24 weeks post-baseline
Change from baseline in ALT | 48 weeks
  Change from baseline in ALT at 48 weeks post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jun Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided